CLINICAL TRIAL: NCT05888337
Title: Comparison of Contoura Vision Outcomes Programmed Using the Manifest Refraction Verses Using Phorcides Planning Software in Patients With Oblique Astigmatism
Status: Terminated | Type: Observational
Why Stopped: Difficult to find recruit patients with oblique astigmatism
Sponsor: Bismarck Lasik (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: SW-23-01
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Contoura LASIK with Phorcides planning strategy
  Interventions: Device: Contoura LASIK with Phorcides planning strategy
- Contoura LASIK with manifest refraction planning strategy
  Interventions: Device: Contoura LASIK with manifest refraction planning strategy

INTERVENTIONS:
Device: Contoura LASIK with Phorcides planning strategy — Bilateral treatment with topography guided LASIK
  Groups: Contoura LASIK with Phorcides planning strategy
Device: Contoura LASIK with manifest refraction planning strategy — Bilateral treatment with topography guided LASIK
  Groups: Contoura LASIK with manifest refraction planning strategy

SUMMARY:
The objective is to compare the percentage of monocular UDVA -0.1 logMAR (20/16) outcomes for each planning strategy (Phorcides and manifest refraction) at the 3-month post operative visit.

DETAILED DESCRIPTION:
This study is a randomized, prospective contralateral eye study of visual outcomes in eyes planned with Phorcides compared to eyes planned using the manifest refraction after successful bilateral LASIK surgery. Subjects will be assessed pre-operatively, operatively and at 3 months postoperatively. Clinical evaluations will include measurement of visual acuity, manifest refraction, and administration of a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above
* Preoperative total corneal Pachymetry 490um or above
* BCVA 20/20 or better
* Stable refractive error <0.50D MRSE change in preceding year
* Good general and ocular health
* Preoperative exam completed within three months of surgery
* Soft contact lens wear discontinued 3 days prior to preoperative exam and the procedure
* Residual stromal bed greater than 270um
* Candidates who qualify for Contoura treatment OU (≤ -8.0 D SPH and ≤ -3.0 D CYL)
* Candidates who elect to target both eyes targeted for emmetropia
* ≤ -3.0 D Oblique astigmatism as defined as an axis between 30-60 degrees or between 120-150 degrees

Exclusion Criteria:

* Subjects with usual relative and absolute contraindications for LASIK surgery (subjects with severe dry eye, subjects with recurrent corneal erosion, subjects with uncontrolled Glaucoma, subjects with collagen vascular disorders, keratoconus or signs of keratoconus, Uncontrolled Diabetes, Herpes, corneal dystrophies or degeneration; any irregular astigmatism)
* Pachymetry below 490
* Autoimmune or immunodeficiency diseases, Pregnant or nursing women
* Subjects with signs of inability to understand consent for study and procedure planned
* Subjects with history of previous ocular surgery

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years of age or older who are interested in and appropriate candidates for LASIK.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Percentage of eyes with monocular UDVA of logMAR -0.10 (20/16) in each group | 3 months postoperatively

SECONDARY OUTCOMES:
Percentage of eyes with monocular UDVA of logMAR -0.20 (20/12.5) in each group | 3 months postoperatively

OTHER OUTCOMES:
Percentage of eyes with monocular UDVA of logMAR 0.00 (20/20) in each group | 3 months postoperatively
Mean/SD of residual refractive error and centroid of manifest refraction (dioptric magnitude of residual astigmatism and residual SE) | 3 months postoperatively
Percentage of eyes with postoperative UDVA equal to or better than their preoperative CDVA | 3 months postoperatively
Percentage of eyes that gained 1 or more lines postoperative CDVA and preoperative CDVA | 3 months postoperatively
Percentage of subjects that report overall visual preference of the Phorcides planned eye vs manifest refraction planned eye | 3 months postoperatively
Quantitative rating of overall satisfaction of vision in each eye | 3 months postoperatively
  Satisfaction will be measured using a questionnaire. Subjects will rate satisfaction with vision in each eye using the scale:
  * Completely Dissatisfied
  * Very Dissatisfied
  * Somewhat Dissatisfied
  * Somewhat Satisfied
  * Very Satisfied
  * Completely Satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Wexler, MD, Principal Investigator — Bismarck Lasik
Locations (1):
- Bismarck Lasik, Bismarck, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No